CLINICAL TRIAL: NCT06706544
Title: Effectiveness and Cost-effectiveness of Ozone Treatment in Patients With Paresthesia (Numbness, Tingling) Secondary to Chemotherapy-induced Peripheral Neuropathy. Randomized, Triple-blind Clinical Trial (OzoParQT)
Brief Title: Ozone Treatment in Paresthesia (Numbness, Tingling) Secondary to Chemotherapy-induced Peripheral Neuropathy
Acronym: OzoParQT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bernardino Clavo, MD, PhD (Other)
Collaborators: Council of Gran Canaria (Other); CIBER (Infectious diseases) (Unknown); Fundacion Canaria Instituto de Investigacion Sanitaria de Canarias (Other); Complejo Hospitalario Universitario Insular Materno Infantil (Other); Servicio de Evaluacion del Servicio Canario de Salud. (Unknown); Institute for Applied Microelectronics, University of Las Palmas de Gran Canaria, Spain (Unknown); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Bernardino Clavo, MD, PhD, Bernardino Clavo, MD, PhD, Dr. Negrin University Hospital, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OzoParQT; PI23/01324 (Other Grant/Funding Number: Instituto de Salud Carlos III); CIGC'23/24 (Other Grant/Funding Number: Cabildo de Gran Canaria); 2024-517196-20-00 (EU CTIS Number); 2023-210-1 (Registry Identifier: CEIm Las Palmas)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN); Paresthesia; Numbness; Tingling
Keywords: Chemotherapy induced peripheral neuropathy; paresthesia; numbness and tingling; side effect of cancer treatment; toxicity of chemotherapy; ozone therapy; quality of life; anxiety; depression; hyperspectral imaging; oxidative stress
MeSH Terms: conditions — Paresthesia; Hypesthesia; Anxiety Disorders; Depression | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: * the oncologists/hematologists who treat and follow the patient regularly,
  * researchers who carry out biochemical determinations or functional tests,
  * the staff who obtain the economic data,
  * statisticians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ozone Group (Experimental): Drug: Ozone (O3/O2). Treatment: Usual treatment + Ozone therapy by rectal insufflation. O3/O2 concentration progressively increased from 10 to 30 μg/ml; 40 sessions in 16 weeks.
  Interventions: Drug: Ozone therapy
- Oxygen Group (Placebo) (Placebo Comparator): Drug: Oxygen (O2). Treatment: Usual treatment + Oxygen by rectal insufflation. O3/O2 concentration = 0 μg/ml (only O2); 40 sessions in 16 weeks.
  Interventions: Drug: Oxygen (placebo)

INTERVENTIONS:
Drug: Ozone therapy — Usual treatment (by their oncologist or hematologist) + Ozone therapy by rectal insufflation. O3/O2 concentration progressively increased from 10 to 30 μg/ml; 40 sessions in 16 weeks.
  Other Names: Ozone treatment; O3; O3/O2 gas mixture
  Arms: Ozone Group
Drug: Oxygen (placebo) — Usual treatment (by their oncologist or hematologist) + Oxygen by rectal insufflation. O3/O2 concentration = 0 μg/ml (only O2); 40 sessions in 16 weeks.
  Other Names: O2
  Arms: Oxygen Group (Placebo)

SUMMARY:
The goal of this phase II/III randomized clinical trial is to evaluate the effect of adding rectal ozone therapy to the usual management of patients with paresthesia (numbness and/or tingling) due to chemotherapy-induced peripheral neuropathy (CIPN). Ozone treatment consists of the rectal insufflation of 180 - 300 milliliters of an ozone/oxygen gas mixture.

The main questions to answer are:

1. Can ozone therapy improve patients' self-perceived level of numbness and tingling?
2. Can ozone therapy improve patients' self-perceived health-related quality of life (HRQoL)?

In 42 patients with chronic numbness and tingling secondary to chemotherapy, the researchers will compare:

* the addition of rectal ozone insufflations
* versus the addition of rectal oxygen insufflations (placebo). Participants will receive 40 rectal gas (ozone versus oxygen) insufflations in 16 weeks and will continue other symptomatic or cancer treatments prescribed by their oncologists.

Before treatment, after treatment, and 12 weeks after treatment, they will be evaluated:

* Several questionnaires about neuropathy, quality of life, and anxiety and depression.
* Biochemical parameters of oxidative stress and inflammation
* Hyperspectral images of hands and feet
* Toxicity of procedure.

DETAILED DESCRIPTION:
Rationale Chemotherapy-induced peripheral neuropathy (CIPN) can lead to a decrease and/or interruption of chemotherapy treatment, limiting its efficacy and decreasing patients' quality of life. Therapeutic measures for CIPN are very limited in number and efficacy. Our previous experience has suggested the potential clinical usefulness of adjuvant treatment with ozone in patients with CIPN. The hypothesis of the trial is that ozone treatment will improve numbness and tingling symptoms in patients with CIPN.

Primary objectives:

To evaluate the effect of adding ozone to the usual management of patients with paresthesia (numbness and/or tingling) due to chemotherapy-induced peripheral neuropathy (CIPN), Grade 2 (moderate symptoms and/or limitation in instrumental activities of daily living) or higher, on:

1. patients' self-perceived level of paresthesia
2. patients' self-perceived health-related quality of life (HRQoL).

Secondary objectives:

To evaluate (in patients with numbness and/or tingling secondary to CIPN) the effect of adding ozone to the usual management on:

1. the additional direct costs incurred in the application of ozone and evaluate the cost-effectiveness of the administration of ozone in these patients in comparison with the usual exclusive treatment.
2. the evolution of the sensory neuropathy
3. the evolution of the level of anxiety and depression,
4. the evolution of biochemical parameters related to oxidative stress and chronic inflammation.
5. the evolution of hyperspectral signatures obtained from hands and feet.
6. to evaluate the toxicity of rectal ozone treatment in these patients.

Main trial endpoints.

1. Percentage of change from baseline in "numbness and tingling" self-perceived by patients at the end of follow-up (week 28 after the commencement of ozone treatment)
2. Change from baseline in "quality of life" (using the EQ-5D-5L questionnaire) self-perceived by patients at the end of follow-up (week 28 after the commencement of ozone treatment)

Secondary trial endpoints.

To evaluate the percentage of change from baseline in all the secondary objectives:

* at the end of ozone treatment (weeks 16)
* and at the end of follow-up (week 28)

Trial design. Phase II-III randomized triple-blind clinical trial. The duration of each patient in the study will be 28 weeks: 16 weeks of treatment and 12 weeks of follow-up. The planned total duration of the project is 60 months.

Trial population. 42 adult patients (>= 18 years old), with any tumor, with paresthesias (numbness and/or tingling) due to CIPN, grade of toxicity >= 2 (according to the Common Toxicity Criteria for Adverse Events (CTCAE) from the National Cancer Institute of EEUU, v.5.0), for >= 3 months.

Intervention.

All patients will receive the usual management and treatment for their symptoms + "40 sessions of rectal insufflation of O3/O2 gas mixture" in 16 weeks (3 or 2 sessions per week):

* Ozone group, O3/O2 concentration increasing from 10 to 30 µg/mL (µg of O3 by mL of O2).
* Control-placebo group, O3/O2 concentration = 0 µg/mL (this is: only O2).

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults > = 18 years old.
* 2. Previous treatment with any chemotherapy because of any tumor.
* 3. Clinical diagnosis of paresthesia (numbness, tingling) secondary to CIPN, with toxicity Grade > = 2 (according to the Common Toxicity Criteria for Adverse Events (CTCAE) from the National Cancer Institute of EEUU, v.5.0) for > = 3 months.
* 4. Without neurotoxic chemotherapy > = 3 months.
* 5. Cancer disease is stable or in remission.
* 6. Life expectancy > = 6 months.
* 7. Before enrollment, women of childbearing potential should obtain a negative result in the serum or urine pregnancy test at the screening visit and accept the use of appropriate contraceptive methods at least from 14 days before the first ozone therapy session up to 14 days after the last one.
* 8. To sign and date the study-specific informed consent

Exclusion Criteria:

* 1. Age < 18 years.
* 2. A woman who is lactating, pregnant, suspected of being pregnant, or a woman of childbearing potential who does not use adequate contraceptive methods.
* 3. Suspected symptoms are due to diabetic or compressive neuropathy.
* 4. Severe psychiatric disorders.
* 5. Inability to complete the quality of life questionnaires.
* 6. Elevation above 5 times the maximum limit of normal creatinine.
* 7. Patient who is hemodynamic or clinically unstable or who requires urgent or short-term interventional measures.
* 8. Neoplasia in progression requiring recent initiation of systemic treatment or maintenance with neurotoxic chemotherapy.
* 9. Life expectancy (for any reason) < 6 months.
* 10. Known allergy to ozone, known glucose 6 phosphate dehydrogenase (G6PD) deficiency, or hemochromatosis.
* 11. Contraindications or impossibility for rectal ozone treatment or to attend regularly to the treatment.
* 12. Not meeting each and every one of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in "numbness and tingling" self-perceived by patients at the end of follow-up (week 28 after the commencement of ozone treatment) | 28 weeks
  Self-reported evaluation of the percentage of "numbness and/or tingling" regarding the basal level. From 100% (basal level, 0% improvement) to 0% (no numbness and tingling, 100% improvement).
Change from Baseline in quality of life by the EQ-... | 28 weeks
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (Best: I have no problem) to 5 (worst: I have an extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analog scale (0 = worst health patient can imagine, 100 = best health patient can imagine).

SECONDARY OUTCOMES:
Direct hospital costs | 28 weeks
  The direct expenses incurred by the hospital in providing services (medication, tests, medical visits…) during the 28 weeks for the study (in euros).
Change from baseline in "numbness and tingling" self-perceived by patients at the end of ozone treatment. | 16
  Self-reported evaluation of the percentage of "numbness and/or tingling" regarding the basal level. From 100% (basal level, 0% improvement) to 0% (no numbness and tingling, 100% improvement).
Changes from baseline in the Grade of toxicity of parestesias (numbness, tingling) according to the CTCAE v.5.0. scale at the end of ozone treatment. | 16 weeks
  Changes from baseline in the Grade of toxicity of paresthesias (numbness, tingling) according to the CTCAE v.5.0. scale (from the National Cancer Institute of EEUU). Range from: Grade = (asymptomatic or mild symptoms) to Grade 3 (severe symptoms, limiting self-care activities in daily life).
Changes from baseline in the Grade of toxicity of sensory neuropathy according to the CTCAE v.5.0. scale at the end of ozone treatment. | 16 weeks.
  Changes from baseline in the Grade of toxicity of paresthesias (numbness, tingling) according to the CTCAE v.5.0. scale (from the National Cancer Institute of EEUU). Range from: Grade = (asymptomatic or mild symptoms) to Grade 4 (life-threatening consequences, urgent intervention indicated).
Changes from baseline in the degree of neuropathy according to the QLQ-CIPN20 scale at the end of ozone treatment. | 16 weeks.
  Changes from baseline in the degree of neuropathy according to the QLQ-CIPN20 scale at the end of ozone treatment (from the European Organization for Research & Treatment in Cancer (EORTC)). It is evaluated through 20 items that are grouped into 3 dimensions: sensitive, motor and autonomic. Range: each item is scored from 1 (nothing) to 4 (a lot). The total score for each dimension is transformed into a score from 0 to 1000, being 0 the best state and 100 the worst.
Change from baseline in "Quality of Life" (using the EQ-5D-5L questionnaire) self-perceived by patients at the end of ozone treatment (week 16 after the commencement of ozone treatment). | 16 weeks.
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (Best: I have no problem) to 5 (worst: I have an extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analog scale (0 = worst health patient can imagine, 100 = best health patient can imagine).
Changes from baseline in the "Quality of Life" according to the QLQ-C30 questionnaire at the end of ozone treatment. | 16 weeks.
  Changes from baseline in the "Quality of Life" according to the QLQ-C30 questionnaire (from the European Organization for Research & Treatment in Cancer (EORTC)). Self-reported evaluation of 30 items that measure several scales and symptoms. Range (after standardization): from 0 (worst for overall health and function, best for symptoms) to 100 (best for overall health and functions, worst for symptoms).
Changes from baseline in levels of anxiety and depression according to the Hospital Anxiety and Depression Scale (HADS), at the end of ozone treatment. | 16 weeks
  Changes from baseline in levels of anxiety and depression according to the Hospital Anxiety and Depression Scale (HADS). HADS is a self-administered questionnaire that assesses 14 items/symptoms of anxiety (7) and depression (7) experienced by patients. Each item is scored from 0 (better, no alteration) to 3 (worse level of alteration). For each symptom (anxiety or depression), the overall score is from 0 (better, no anxiety or depression) to 21 (worse, very severe anxiety or depression).
Changes from baseline in biochemical parameters of oxidative stress at the end of ozone treatment. | 16 weeks.
  Changes in serum levels of superoxide dismutase, glutathione, glutathione peroxidase and free radicals
Changes from baseline in biochemical parameters of inflammation at the end of ozone treatment. | 16 weeks
  Changes in serum levels of pro-inflammatory cytokines.
Changes from baseline in Hyperspectral signatures and infrared images obtained from hands and feet at then of ozone treatment. | 16 weeks
  Assessment of the percentage of reflectance for each wavelength of the hyperspectral and infrared images obtained with specific devices.
Changes from baseline in the Grade of toxicity of paresthesias (numbness, tingling) according to the CTCAE v.5.0. scale at the end of follow-up. | 28 weeks.
  Changes from baseline in the Grade of toxicity of paresthesias (numbness, tingling) according to the CTCAE v.5.0. scale (from the National Cancer Institute of EEUU). Range from: Grade = (asymptomatic or mild symptoms) to Grade 3 (severe symptoms, limiting self-care activities in daily life).
Changes from baseline in the Grade of toxicity of sensory neuropathy according to the CTCAE v.5.0. scale at the end of follow-up. | 28 weeks
  Changes from baseline in the Grade of toxicity of paresthesias (numbness, tingling) according to the CTCAE v.5.0. scale (from the National Cancer Institute of EEUU). Range from: Grade = (asymptomatic or mild symptoms) to Grade 4 (life-threatening consequences, urgent intervention indicated).
Changes from baseline in the degree of neuropathy according to the QLQ-CIPN20 scale at the end of follow-up. | Time frame: 28 weeks
  Changes from baseline in the degree of neuropathy according to the QLQ-CIPN20 scale at the end of ozone treatment (from the European Organization for Research & Treatment in Cancer (EORTC)). It is evaluated through 20 items that are grouped into 3 dimensions: sensitive, motor, and autonomic. Range: each item is scored from 1 (nothing) to 4 (a lot). The total score for each dimension is transformed into a score from 0 to 1000, being 0 the best state and 100 the worst.
Changes from baseline in the "Quality of Life" according to the QLQ-C30 questionnaire at the end of follow-up. | 28 weeks.
  Changes from baseline in the "Quality of Life" according to the QLQ-C30 questionnaire (from the European Organization for Research & Treatment in Cancer (EORTC)). Self-reported evaluation of 30 items that measure several scales and symptoms. Range (after standardization): from 0 (worst for overall health and function, best for symptoms) to 100 (best for overall health and functions, worst for symptoms).
Changes from baseline in levels of anxiety and depression according to the Hospital Anxiety and Depression Scale (HADS) at the end of follow-up. | 28 weeks.
  Changes from baseline in levels of anxiety and depression according to the Hospital Anxiety and Depression Scale (HADS). HADS is a self-administered questionnaire that assesses 14 items/symptoms of anxiety (7) and depression (7) experienced by patients. Each item is scored from 0 (better, no alteration) to 3 (worse level of alteration). For each symptom (anxiety or depression), the overall score is from 0 (better, no anxiety or depression) to 21 (worse, very severe anxiety or depression).
Changes from baseline in biochemical parameters of oxidative stress at the end of follow-up. | 28 weeks.
  Changes in serum levels of superoxide dismutase, glutathione, glutathione peroxidase and free radicals.
Changes from baseline in biochemical parameters of inflammation at the end of follow-up. | 28 weeks.
  Changes in serum levels of pro-inflammatory cytokines.
Changes from baseline in Hyperspectral signatures and infrared images obtained from hands and feet at the end of follow-up. | 28 weeks.
  Assessment of the percentage of reflectance for each wavelength of the hyperspectral and infrared images obtained with specific devices.
Toxicity of rectal ozone treatment at the end of follow-up. | 28 weeks.
  Grade of toxicity secondary to the rectal insufflation of the rectal ozone treatment according to the CTCAE v.5.0. scale (from the National Cancer Institute of EEUU).

CONTACTS AND LOCATIONS:
Overall Officials: Bernardino Clavo, MD, PhD, Study Chair — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain; Francisco Rodríguez-Esparragón, BSc, PhD, Study Director — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain; Himar Fabelo, BSc, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain; Gustavo M Callicó, Prof, PhD, Principal Investigator — Institute for Applied Microelectronics, University of Las Palmas de Gran Canaria, Spain; Francisco Rodríguez-Esparragón, BSc, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain; Bernardino Clavo, MD, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain
Locations (1):
- Dr. Negrín University Hospital, Las Palmas, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Yes
It will be available (after request):
  * Individual participant data (IPD) that underlie the results reported in further articles, after deidentification
  * Data will be available after publication, ending 36 months following article publication.
  * They will be available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  * Study protocol
  Proposals should be directed to: bernardinoclavo@gmail.com To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after publication, ending 36 months following article publication.
Access Criteria: Data will be available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  - Study protocol
  Proposals should be directed to: bernardinoclavo@gmail.com To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Viebahn-Haensler R, Leon Fernandez OS. Ozone in Medicine. The Low-Dose Ozone Concept and Its Basic Biochemical Mechanisms of Action in Chronic Inflammatory Diseases. Int J Mol Sci. 2021 Jul 23;22(15):7890. doi: 10.3390/ijms22157890. PMID 34360655
- [Background] Tricarico G, Travagli V. The Relationship between Ozone and Human Blood in the Course of a Well-Controlled, Mild, and Transitory Oxidative Eustress. Antioxidants (Basel). 2021 Dec 4;10(12):1946. doi: 10.3390/antiox10121946. PMID 34943049
- [Background] Szklener K, Rudzinska A, Juchaniuk P, Kabala Z, Mandziuk S. Ozone in Chemotherapy-Induced Peripheral Neuropathy-Current State of Art, Possibilities, and Perspectives. Int J Mol Sci. 2023 Mar 9;24(6):5279. doi: 10.3390/ijms24065279. PMID 36982352
- [Background] Smith EM, Pang H, Cirrincione C, Fleishman S, Paskett ED, Ahles T, Bressler LR, Fadul CE, Knox C, Le-Lindqwister N, Gilman PB, Shapiro CL; Alliance for Clinical Trials in Oncology. Effect of duloxetine on pain, function, and quality of life among patients with chemotherapy-induced painful peripheral neuropathy: a randomized clinical trial. JAMA. 2013 Apr 3;309(13):1359-67. doi: 10.1001/jama.2013.2813. PMID 23549581
- [Background] Hidalgo-Tallon J, Menendez-Cepero S, Vilchez JS, Rodriguez-Lopez CM, Calandre EP. Ozone therapy as add-on treatment in fibromyalgia management by rectal insufflation: an open-label pilot study. J Altern Complement Med. 2013 Mar;19(3):238-42. doi: 10.1089/acm.2011.0739. Epub 2012 Oct 9. PMID 23046293
- [Background] Hidalgo-Tallon FJ, Torres-Morera LM, Baeza-Noci J, Carrillo-Izquierdo MD, Pinto-Bonilla R. Updated Review on Ozone Therapy in Pain Medicine. Front Physiol. 2022 Feb 23;13:840623. doi: 10.3389/fphys.2022.840623. eCollection 2022. PMID 35283802
- [Background] Galie M, Covi V, Tabaracci G, Malatesta M. The Role of Nrf2 in the Antioxidant Cellular Response to Medical Ozone Exposure. Int J Mol Sci. 2019 Aug 17;20(16):4009. doi: 10.3390/ijms20164009. PMID 31426459
- [Background] Clavo B, Suarez G, Aguilar Y, Gutierrez D, Ponce P, Cubero A, Robaina F, Carreras JL. Brain ischemia and hypometabolism treated by ozone therapy. Forsch Komplementmed. 2011;18(5):283-7. doi: 10.1159/000333795. Epub 2011 Oct 13. PMID 22105041
- [Background] Clavo B, Rodriguez-Esparragon F, Rodriguez-Abreu D, Martinez-Sanchez G, Llontop P, Aguiar-Bujanda D, Fernandez-Perez L, Santana-Rodriguez N. Modulation of Oxidative Stress by Ozone Therapy in the Prevention and Treatment of Chemotherapy-Induced Toxicity: Review and Prospects. Antioxidants (Basel). 2019 Nov 26;8(12):588. doi: 10.3390/antiox8120588. PMID 31779159
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Long-Term Results with Adjuvant Ozone Therapy in the Management of Chronic Pelvic Pain Secondary to Cancer Treatment. Pain Med. 2021 Sep 8;22(9):2138-2141. doi: 10.1093/pm/pnaa459. No abstract available. PMID 33738491
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Ozone Therapy in Refractory Pelvic Pain Syndromes Secondary to Cancer Treatment: A New Approach Warranting Exploration. J Palliat Med. 2021 Jan;24(1):97-102. doi: 10.1089/jpm.2019.0597. Epub 2020 May 5. PMID 32379556
- [Background] Clavo B, Rodriguez-Abreu D, Galvan S, Federico M, Martinez-Sanchez G, Ramallo-Farina Y, Antonelli C, Benitez G, Rey-Baltar D, Jorge IJ, Rodriguez-Esparragon F, Serrano-Aguilar P. Long-term improvement by ozone treatment in chronic pain secondary to chemotherapy-induced peripheral neuropathy: A preliminary report. Front Physiol. 2022 Aug 30;13:935269. doi: 10.3389/fphys.2022.935269. eCollection 2022. PMID 36111149
- [Background] Clavo B, Martinez-Sanchez G, Rodriguez-Esparragon F, Rodriguez-Abreu D, Galvan S, Aguiar-Bujanda D, Diaz-Garrido JA, Canas S, Torres-Mata LB, Fabelo H, Tellez T, Santana-Rodriguez N, Fernandez-Perez L, Marrero-Callico G. Modulation by Ozone Therapy of Oxidative Stress in Chemotherapy-Induced Peripheral Neuropathy: The Background for a Randomized Clinical Trial. Int J Mol Sci. 2021 Mar 10;22(6):2802. doi: 10.3390/ijms22062802. PMID 33802143
- [Background] Clavo B, Ceballos D, Gutierrez D, Rovira G, Suarez G, Lopez L, Pinar B, Cabezon A, Morales V, Oliva E, Fiuza D, Santana-Rodriguez N. Long-term control of refractory hemorrhagic radiation proctitis with ozone therapy. J Pain Symptom Manage. 2013 Jul;46(1):106-12. doi: 10.1016/j.jpainsymman.2012.06.017. Epub 2012 Oct 26. PMID 23102757
- [Background] Clavo B, Canovas-Molina A, Ramallo-Farina Y, Federico M, Rodriguez-Abreu D, Galvan S, Ribeiro I, Marques da Silva SC, Navarro M, Gonzalez-Beltran D, Diaz-Garrido JA, Cazorla-Rivero S, Rodriguez-Esparragon F, Serrano-Aguilar P. Effects of Ozone Treatment on Health-Related Quality of Life and Toxicity Induced by Radiotherapy and Chemotherapy in Symptomatic Cancer Survivors. Int J Environ Res Public Health. 2023 Jan 13;20(2):1479. doi: 10.3390/ijerph20021479. PMID 36674232
- [Background] Clavo B, Canovas-Molina A, Diaz-Garrido JA, Canas S, Ramallo-Farina Y, Laffite H, Federico M, Rodriguez-Abreu D, Galvan S, Garcia-Lourve C, Gonzalez-Beltran D, Carames MA, Hernandez-Fleta JL, Serrano-Aguilar P, Rodriguez-Esparragon F. Effects of ozone therapy on anxiety and depression in patients with refractory symptoms of severe diseases: a pilot study. Front Psychol. 2023 Aug 4;14:1176204. doi: 10.3389/fpsyg.2023.1176204. eCollection 2023. PMID 37599784
- [Background] Bocci VA, Zanardi I, Travagli V. Ozone acting on human blood yields a hormetic dose-response relationship. J Transl Med. 2011 May 17;9:66. doi: 10.1186/1479-5876-9-66. PMID 21575276
- [Background] Bocci V, Valacchi G. Nrf2 activation as target to implement therapeutic treatments. Front Chem. 2015 Feb 2;3:4. doi: 10.3389/fchem.2015.00004. eCollection 2015. PMID 25699252
- [Background] Bocci V, Borrelli E, Travagli V, Zanardi I. The ozone paradox: ozone is a strong oxidant as well as a medical drug. Med Res Rev. 2009 Jul;29(4):646-82. doi: 10.1002/med.20150. PMID 19260079